CLINICAL TRIAL: NCT02129309
Title: Haemodynamic Effects of Apelin Agonists and Antagonists in Man in COPD With Raised Pulmonary Artery Pressures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Wellcome Trust (Other); University of Cambridge (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Physician & Clinical Pharmacologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ALPHa-COPD
Record Dates: First submitted 2014-04-28; First posted 2014-05-02 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-01

CONDITIONS: COPD; Pulmonary Hypertension
Keywords: COPD; Apelin; agonist; antagonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systemic Apelin infusion (Experimental): Study 2a - Haemodynamic studies to investigate the response to systemic infusions of 3 apelin agonists in healthy volunteers
  Study 2b - Haemodynamic studies to investigate the response to 3 apelin agonists in COPD patients with elevated pulmonary artery pressures
  Interventions: Procedure: Haemodynamic studies
- Apelin infusion - forearm (Experimental): Study 1a - A validation dose study of 3 apelin agonists using forearm plethysmography to evaluate changes in forearm blood flow: performed in healthy volunteers and COPD patients with elevated pulmonary artery pressures.
  Study 1b- A validation dose study of apelin receptor antagonist using forearm plethysmography to evaluate changes in forearm blood flow, in healthy volunteers and COPD patients with elevated pulmonary artery pressures.
  Interventions: Procedure: Forearm plethysmography

INTERVENTIONS:
Procedure: Forearm plethysmography — Dose response study
  Arms: Apelin infusion - forearm
Procedure: Haemodynamic studies — Dose response study
  Other Names: Innocor; Bioimpedance; Echocardiography
  Arms: Systemic Apelin infusion

SUMMARY:
The investigators are interested in studying how Pulmonary Hypertension occurs. A substance called 'apelin', that naturally occurs in the body has been shown to have an important role in heart disease. Previous studies have shown that it can make blood vessels get wider, and help blood flow around the body and thus improve the way the heart and lungs work.

The investigators are looking to recruit both healthy and COPD pulmonary hypertension patients to study 3 types of apelin. The purpose of this study is to help the investigators understand how Pulmonary Hypertension occurs which may will help with the development of future treatments.

DETAILED DESCRIPTION:
The purpose of this study:

To investigate the physiological role of apelin in the cardiovascular system in patients with COPD with raised pulmonary artery pressures.

Study Aim and hypotheses:

The primary objective is to test the above hypotheses using forearm blood flow and systemic infusions of apelin peptides.

Hypotheses:

1. Apelin agonists are vasodilators in human resistance vessels and this effect will be altered in patients with pulmonary hypertension.
2. Apelin peptides improve right ventricular and pulmonary haemodynamics in patients with elevated pulmonary artery pressures.

Study 1a - A validation dose study of 3 apelin agonists performed in healthy volunteers and COPD patients with elevated pulmonary artery pressures.

Study 1b- A validation dose study of apelin receptor antagonist, in healthy volunteers and COPD patients with elevated pulmonary artery pressures.

Study 2a - To define the haemodynamic response to apelin agonists in healthy volunteers and evaluate the response.

Study 2b - To investigate the haemodynamic response to 3 apelin agonists in COPD patients with elevated pulmonary artery pressures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

  * Aged 18 to 70 years
  * Non-smoker (<1 cigarette per week)
  * If female, postmenopausal or on days 2-9 of menstrual cycle and negative pregnancy test COPD patients with estimated Pulmonary Artery Pressure (PAP) on echo >25mmHg
  * Clinical diagnosis of COPD as per standard criteria
  * Between 18 and 70 years
  * If female, postmenopausal or on days 2-9 of menstrual cycle and negative pregnancy test

Exclusion Criteria:

* pre-existing:

  * Systemic Hypertension (sustained BP >160/100mmHg)
  * Ischaemic Heart Disease
  * Primary valvular heart disease
  * Significant left ventricular failure
  * Active malignancy
  * Renal disease (Creatinine >180 µmol/L)
  * Neurological disease
  * Diabetes mellitus
  * BMI >35, BMI <17
  * Pregnancy
  * Use of vasoactive medication or NSAIDS/aspirin within 48 hours of study.
  * Current involvement in other research studies, other than observational/non-interventional
  * Known HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage change in forearm blood flow in the infused arm. Forearm blood flow ratio in each arm, blood pressure and heart rate will also be reported. | 12 months
Cardiac output and stroke volume, pulmonary vascular resistance, mean arterial pressure and heart rate. | 12 months

OTHER OUTCOMES:
Exploratory endpoints in Study 2 are systolic and diastolic blood pressure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joseph Cheriyan, MD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Vascular Research Unit, Clinical Pharmacology Unit, ACCI, Level 3, Addenbrooke's Hospital, Hills Road, Cambridge, United Kingdom